CLINICAL TRIAL: NCT05886946
Title: Arterial Blood Gas as an Early Screening Tool for Predicting Lung Injury in Blunt Chest Trauma
Brief Title: Abg in Blunt Chest Trauma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, asmaa ali mohamed hasan, Assistant lecturer, Assiut University
Other Study IDs: Abg in blunt chest
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2022-12

CONDITIONS: Blunt Injury of Thorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ABG — ABG

SUMMARY:
This study aims to determine the value of ABG measurments in patients with blunt chest trauma and its role in prognosis of different outcomes and the results would aid the emergency physicians to speed up the management and reduce the cost of diagnosis

ELIGIBILITY:
Inclusion Criteria:

- all patient with polytrauma or blunt trauma to chest and thoraco-abdominal area from both genders are included in the study

Exclusion Criteria:

* shocked patients whom were intubated ,patients that had pulmonary disease or heart diseases ,penetrating chest injury ,pregnant female ,patients who do not want to participate in the study

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: blunt chest trauma
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Arterial blood gas as an early screening tool for predicting lung injury in blunt chest trauma | 5 minutes after arrival to emergency
  evaluate the diagnostic accuracy of ABG as a screening tool for identifying and early diagnosis lung injury in adult in blunt chest trauma

IPD SHARING:
Plan to Share IPD: Undecided
no plain now